CLINICAL TRIAL: NCT04581330
Title: The Effects of Fractional CO2 Laser on Poikiloderma of Civatte
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Heather Woodworth Goff, Primary Investigator, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: STU-2020-0827
Record Dates: First submitted 2020-10-02; First posted 2020-10-09 (Actual); Results first posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-02

CONDITIONS: Poikiloderma of Civatte

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- DEKA SmartXide C02 laser (Experimental): One half of the subject's neck will be treated with ablative fractional CO2 laser.
  Interventions: Device: DEKA SmartXide C02 laser
- Control (No Intervention): The other half of the subject's neck will not be treated with the ablative fractional CO2 laser.

INTERVENTIONS:
Device: DEKA SmartXide C02 laser — One pass with a 1-mm spot density and a 60 micron depth will be performed followed by a 1-mm spot density and a 200 micron depth will be used
  Arms: DEKA SmartXide C02 laser

SUMMARY:
This study will assess the safety and efficacy of fractional CO2 laser treatment for Poikiloderma of Civatte (POC).POC is a chronic vascular and pigmentary disorder typically involving the lateral and inferior neck region, as well as the chest area. Clinically, poikiloderma appears as a combination of telangiectasia, irregular pigmentation, and atrophic changes.Little data exist regarding the use of fractional CO2 laser for management of POC. This study hopes to fulfill this purpose. The primary outcome will be a blinded assessment by dermatologists in the improvement in POC using the Physician's Global Aesthetic Improvement Scale following therapy. The secondary outcomes include subject satisfaction post-treatment and assessment of all procedure-related adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, English and non-English speakers, and subjects more than 18 years old
* Clinical diagnosis of poikiloderma of Civatte affecting the neck and chest
* Agree to not undergo any other procedures on the neck and chest area during the study
* Agree to refrain from tanning for 6 months post-procedure
* Willing and able to read, understand, and sign the consent form
* Willing and able to adhere to the treatment and follow-up schedule as well as post-treatment care

Exclusion Criteria:

* Patients under 18 years old
* Active skin infection, dermatitis, or a rash on the treatment area
* Pregnant or lactating patients
* Patients on immunosuppressive medications
* Any laser procedures or chemical peel procedures on the neck or chest area within the past 6 months
* Patients with multiple comorbidities such as diabetes mellitus, cardiovascular diseases, neurologic disorders, internal malignancies
* Personal history or family history of forming keloids or hypertrophic scars, or abnormal wound healing
* Patients with known bleeding disorders or taking more than one anticoagulation medications
* Undergoing any surgery in the treatment area within the past 12 months
* History of radiation to the head, neck, and chest area
* Systemic use of isotretinoin within 6 months
* Any use of gold therapy
* Current smoker or history of smoking within 12 months of study
* Any physical or mental condition in which the investigators deem unsafe for the subject to participate in the study.
* History of recurrent herpes simplex on the neck or chest.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather W Goff, MD, Principal Investigator — University of Texas at Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- [Background] Katoulis AC, Stavrianeas NG, Georgala S, Bozi E, Kalogeromitros D, Koumantaki E, Katsambas AD. Poikiloderma of Civatte: a clinical and epidemiological study. J Eur Acad Dermatol Venereol. 2005 Jul;19(4):444-8. doi: 10.1111/j.1468-3083.2005.01213.x. PMID 15987290

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The Control Arm assignment consists of the same participants from the intervention arm, but the only difference is that the other half of the participant's neck was considered as the Control which was not treated with the ablative fractional CO2 laser.
Units Other Than Participants: side of the neck
Groups:
- Control: No Intervention: The other half of the subject's neck will not be treated with the ablative fractional CO2 laser.
Period: Overall Study
Arm/Group | DEKA SmartXide C02 Laser | Control
Started | 10; 10 side of the neck | 10; 10 side of the neck
Completed | 10; 10 side of the neck | 10; 10 side of the neck
Not Completed | 0; 0 side of the neck | 0; 0 side of the neck

BASELINE CHARACTERISTICS:
Population: The Control Arm assignment consists of the same participants from the intervention arm, but the only difference is that the other half of the participant's neck was considered as the Control which was not treated with the ablative fractional CO2 laser.
Groups:
- All Participants: One half of the subject's neck will be treated with ablative fractional CO2 laser (DEKA SmartXide ).
  One pass with a 1-mm spot density and a 60 micron depth will be performed followed by a 1-mm spot density and a 200 micron depth will be used.
  The other half of the subject's neck will not be treated with the ablative fractional CO2 laser.
Arm/Group | All Participants
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Overall Improvement of Poikiloderma of Civatte (POC) From Baseline at 12 Weeks
Description: Improvement of Poikiloderma of Civatte (POC) at 12 weeks post treatment is assessed by the Physician's Global Aesthetic Improvement Scale which is a 10-point scale. Each dermatologist from an independent panel (blinded to treatment parameters and the treatment laterality at each photograph time point) will be asked to identify the baseline and post-treatment images from randomized, paired images for all subjects. Reviewers will rate improvement of POC in 10% increments on a 10-point scale (0% no improvement to 100% or complete clearance).
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: percentage
Units Other Than Participants: side of the neck
Arm/Group | DEKA SmartXide C02 Laser | Control
Number analyzed (Participants) | 10 | 10
Number analyzed (side of the neck) | 10 | 10
percentage
  Improvement in Dyschromia | 11.01 (14.91) | 6.03 (11.94)
  Improvement in Texture | 8.51 (12.69) | 5.89 (10.50)
  Lack of Erythema | 4.33 (13.68) | 2.49 (11.99)

2. Primary Outcome: Change in Overall Improvement of Poikiloderma of Civatte (POC) From Baseline at 24 Weeks
Description: Improvement of Poikiloderma of Civatte (POC) at 24 weeks post treatment is assessed by the Physician's Global Aesthetic Improvement Scale which is a 10-point scale. Each dermatologist from an independent panel (blinded to treatment parameters and the treatment laterality at each photograph time point) will be asked to identify the baseline and post-treatment images from randomized, paired images for all subjects. Reviewers will rate improvement of POC in 10% increments on a 10-point scale (0% no improvement to 100% or complete clearance)
Time Frame: Baseline, 24 weeks post-treatment
Population: Data were not collected because the plan of doing this assessment was dropped due to the COVID-19 pandemic.
Units Other Than Participants: side of the neck
Arm/Group | DEKA SmartXide C02 Laser | Control
Number analyzed (Participants) | 0 | 0
Number analyzed (side of the neck) | 0 | 0

3. Secondary Outcome: Patient Satisfaction Assessment Scores at 12 Weeks Post Treatment
Description: Subjects will assess satisfaction with change of POC using the Global Aesthetic Improvement Scale which is a 5-point satisfaction scale. Scale ranges from 1 to 5, lower score indicating lower satisfaction.
Time Frame: 12 weeks post-treatment
Population: The Control Arm assignment consists of the same participants from the intervention arm, but the only difference is that the other half of the participant's neck was considered as the Control which was not treated with the ablative fractional CO2 laser. Hence satisfaction assessment was done only once with this set of participants and no data available to report in the Control arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DEKA SmartXide C02 Laser | Control
Number analyzed (Participants) | 10 | 0
score on a scale | 4.5 (0.53) |

4. Secondary Outcome: Patient Satisfaction Assessment Scores at 24 Weeks Post Treatment
Description: as for outcome 3
Time Frame: 24 weeks post-treatment
Population: Data were not collected because the plan of doing this assessment was dropped due to the COVID-19 pandemic.
Arm/Group | DEKA SmartXide C02 Laser | Control
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of at Least One Procedure-related Adverse Events
Description: Number of at least one procedure-related adverse events >=Grade 3, as defined by Common Terminology Criteria for Adverse Events by CTCAE v4.0
Time Frame: 24 weeks post-laser treatment
Population: The Control Arm consists of the same participants from the intervention arm, but the only difference is that the other half of the participant's neck was considered as the Control which was not treated with the ablative fractional CO2 laser.
Measure: Number; unit: events
Units Other Than Participants: side of the neck
Groups:
- Control: No Intervention was involved in the Control Arm since the other half of the subject's neck was considered as the Control which was not treated with the ablative fractional CO2 laser
Arm/Group | DEKA SmartXide C02 Laser | Control
Number analyzed (Participants) | 10 | 10
Number analyzed (side of the neck) | 10 | 10
events | 0 | 0

ADVERSE EVENTS:
Time Frame: From Baseline up to 6 months post-treatment
Description: The Control Arm consists of the same participants from the intervention arm, but the only difference is that the other half of the participant's neck was considered as the Control which was not treated with the ablative fractional CO2 laser compared to the other side of the neck which underwent intervention. The unit of assignment is "side of the neck" for each arm.
Arm/Group | DEKA SmartXide C02 Laser | Control
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-09): https://cdn.clinicaltrials.gov/large-docs/30/NCT04581330/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-09): https://cdn.clinicaltrials.gov/large-docs/30/NCT04581330/ICF_001.pdf